CLINICAL TRIAL: NCT05288868
Title: The Effect of Simulation-based Training on Confidence and Competence in Obtaining Vitals in a Child With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-05023509
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Intervention: online didactic lecture and educational simulation activity (Experimental): The didactic was created by the research team and provides information on Autism Spectrum Disorder (ASD) and an approach to taking vital signs in these children. The didactic will be pre-recorded and sent by email to employee study participants. The didactic will last about 10 minutes.
  The simulation activity will have the premise of a child with ASD and their caregiver at clinic visit. The employee participant will be asked to take vital signs on the patient. The caregiver will be played by an actor and the child will be played by a mannequin. An iterative script will be used by the actor during the scenario. The simulation will last about 20 minutes and will be followed by a 10 minute debrief.
  Interventions: Other: Educational Intervention: online didactic lecture and educational simulation activity
- Caregiver Satisfaction (No Intervention): Caregivers who accompany their children with autism to the clinic will be surveyed for their comfort scores before and after the study participants' educational intervention

INTERVENTIONS:
Other: Educational Intervention: online didactic lecture and educational simulation activity — The didactic was created by the research team and provides information on Autism Spectrum Disorder (ASD) and an approach to taking vital signs in these children. The didactic will be pre-recorded and sent by email to employee study participants. The didactic will last about 10 minutes.
  The simulation activity will have the premise of a child with ASD and their caregiver at clinic visit. The employee participant will be asked to take vital signs on the patient. The caregiver will be played by an actor and the child will be played by a mannequin. An iterative script will be used by the actor during the scenario. The simulation will last about 20 minutes and will be followed by a 10 minute debrief.
  Arms: Educational Intervention: online didactic lecture and educational simulation activity

SUMMARY:
The objective is to evaluate the efficacy of an online learning module combined with high fidelity simulation-based training in improving medical assistants' and registered nurses' self-confidence and competence scores in taking vital signs in a child with Autism Spectrum Disorder in clinic. The study will explore the efficacy of high-fidelity simulation which has not been studied to date as a training modality for teaching healthcare workers about Autism Spectrum Disorder. The investigators will also evaluate patient encounter data to provide insight into trainees' transformation of knowledge into clinical practice. The hypothesis is that nurses and medical assistants who participate in an online learning module combined with simulation-based training will demonstrate improved self-confidence and competence scores in evaluating children with Autism.

DETAILED DESCRIPTION:
The study is an interrupted time series design trial. The employee participants will undergo two educational interventions: an online didactic lecture and an educational simulation activity. These activities are both standard educational activities. The online didactic lecture will be recorded and viewed by the participant within a two-week time frame. The simulation activity will be completed in a clinic room in Helmsley Tower 3 or 5 which is an accepted WCM educational setting. An iterative script will be used for the simulation.

The recruitment period for primary study population will last 4 weeks (Week 0 - Week 4).

During this period employee participants will be emailed the study invitation letter, consent form, and survey. A roster of participant names and email addresses will be collected from the consent forms and used throughout the study to email study participants to complete the surveys and participate in the educational interventions. At the start of Week 4 the employee participants will be emailed an online didactic lecture on taking vital signs in children with ASD and they will have 2 weeks to complete the lecture. At the start of Week 9 the employees will be emailed a second survey (post-didactic survey) and will have

1 week to complete it. Prior to week 10 the participants will be emailed to set up a time for their simulation. Then, between Weeks 10-12 they will participate in a simulation activity.

At the start of Weeks 15 the participants will be emailed the final survey (post-simulation survey) which they will have 1 week to complete.

The employee survey will be completed on RedCap and consist of knowledge assessment questions and self-assessment questions.

Parent/guardian surveys will be administered and collected throughout the duration of the study (16 weeks). The parent/guardian surveys will be completed through RedCap or on paper. All surveys completed on paper will not ask for identifying information. A consent document will be provided to participants but will not require a signature for parents electing to complete the survey anonymously on paper. All surveys completed through RedCap will include questions that have identifying information and informed consent will be obtained for participants enrolling in this part of the study. Both the paper and RedCap surveys for guardians will consist of questions inquiring about prior difficulties their child had when having vitals taken, the degree of distress of their child while vital signs were taken during this encounter, strategies the nurse or medical assistant used to approach taking vital signs, and how helpful the strategies were. The number or vital signs obtained during the visit and the duration of time from check-in to rooming will be collected from patient chart review. The patient data will not be linked to data collected from the nurses and medical assistants or to nurses or medical assistants involved in the encounter.

The didactic was created by the research team and provides information on Autism Spectrum Disorder and an approach to taking vital signs in these children. The didactic will be pre-recorded and sent by email to employee study participants. The didactic will last about 10 minutes.

The simulation activity will have the premise of a child with ASD and their caregiver at clinic visit. The employee participant will be asked to take vital signs on the patient. The caregiver will be played by an actor and the child will be played by a mannequin. An iterative script will be used by the actor during the scenario. The simulation will last about 20 minutes and will be followed by a 10 minute debrief.

ELIGIBILITY:
Inclusion Criteria:

* [Primary study participants] any nurses and medical assistants employed in the pediatric clinics of HT3 and HT5.
* [Secondary study participants] pediatric patients ages 1-17 years in HT3 and HT5 clinics with autism spectrum disorder who need vital signs obtained, accompanied by a parent or guardian who can read, write and understand written English.

Exclusion Criteria:

* [Primary study participants] persons who are not nurses or medical assistants employed in the pediatric clinics of HT3 and HT5.
* [Secondary study participants] any patients who do not have a diagnosis of Autism Spectrum Disorder documented in the medical record, are not between the ages of 1 and 17, do not need vital signs obtained at their visit, or are not accompanied by a parent/guardian who can read, write and understand written English.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in confidence scores on the employee questionnaire at weeks 10 and 16 | 0 weeks = baseline; 10 weeks = interim survey; 16 weeks = final survey
  Minimum score = 3 (least confident). Maximum score = 15 (most confident).
Mean change from baseline in competency scores on the employee questionnaire at weeks 10 and 16 | 0 weeks = baseline; 10 weeks = interim survey; 16 weeks = final survey
  Minimum score = 8 (least competent). Maximum score = 40 (most competent).

SECONDARY OUTCOMES:
Mean change from baseline in knowledge scores on the employee questionnaire at weeks 10 and 16 | 0 weeks = baseline; 10 weeks = interim survey; 16 weeks = final survey
  Minimum score = 0 (least knowledgeable); Maximum score = 7 (most knowledgeable)
Mean change from baseline in caregiver satisfaction score on the caregiver survey between weeks 6-10 and 12-16 | 0 weeks = baseline; 6-10 weeks = interim survey; 12-16 weeks = final survey
  Least satisfied = 5. Most satisfied = 1.
Mean change in the number of times vital signs obtained between weeks 0-4, weeks 6-10, and weeks 12-16 | 0 weeks = baseline; 6-10 weeks = interim survey; 12-16 weeks = final survey
  Maximum # of times vital signs obtained = unknown. Minimum # of times vital signs obtained = 1.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Ching, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No